CLINICAL TRIAL: NCT00912964
Title: A Phase III, Randomized, Double-Blind, Parallel Group, Placebo Controlled, Multicenter Study to Assess the Efficacy and Safety of the Beta-3 Agonist Mirabegron (25 mg qd and 50 mg qd) in Subjects With Symptoms of Overactive Bladder
Brief Title: A Study to Test the Efficacy and Safety of the Beta-3 Agonist Mirabegron (YM178) in Patients With Symptoms of Overactive Bladder
Acronym: CAPRICORN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 178-CL-074; 2008-007087-42 (EudraCT Number)
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Results first posted 2012-10-17 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder, Overactive
Keywords: Urgency; YM178; Urinary incontinence; Mirabegron; Micturition; Frequency; Urinary urgency incontinence; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received matching mirabegron placebo tablets orally once a day for 12 weeks.
  Interventions: Drug: Placebo
- Mirabegron 25 mg (Experimental): Participants received mirabegron 25 mg tablets orally once a day for 12 weeks.
  Interventions: Drug: Mirabegron
- Mirabegron 50 mg (Experimental): Participants received mirabegron 50 mg tablets orally once a day for 12 weeks.
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — Mirabegron tablets
  Other Names: YM178; Myrebtriq
  Arms: Mirabegron 25 mg; Mirabegron 50 mg
Drug: Placebo — Matching mirabegron placebo tablets.
  Arms: Placebo

SUMMARY:
The study is intended to test efficacy, safety and tolerability of two doses of once daily (qd) Mirabegron against placebo to treat patients with symptoms of overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to complete the micturition diary and questionnaires correctly
* Patient has symptoms of overactive bladder (OAB) for ≥ 3 months
* Patient must experience frequency of micturition on average ≥ 8 times per 24-hour period during the 3-day micturition diary period
* Patient must experience at least 3 episodes of urgency (grade 3 or 4) with or without incontinence during the 3-day micturition diary period

Exclusion Criteria:

* Patient is breastfeeding, pregnant, intends to become pregnant during the study, or of childbearing potential, sexually active and not practicing a highly reliable method of birth control
* Patient has significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor
* Patient is using medications intended to treat OAB
* Patient has an indwelling catheter or practices intermittent self-catheterization
* Patient has diabetic neuropathy
* Patient has evidence of urinary tract infection, chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs
* Patient receives non-drug treatment including electro-stimulation therapy
* Patient has severe hypertension
* Patient has participated in a clinical study within 30 days, or had participated in any previous study with mirabegron
* Patient had an average total daily urine volume > 3000 mL as recorded in the 3-day micturition diary period
* Patient has serum creatinine of >150 μmol/L, or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2x upper limit of normal range (ULN), or gamma-glutamyl transpeptidase (γ-GT) > 3x ULN
* Patient has a clinically significant abnormal electrocardiogram (ECG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2030 (Actual)
Dates: Start 2009-04-28 (Actual); Primary Completion 2010-04-27 (Actual); Study Completion 2010-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (141):
- United States (78):
  - Homewood, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Chandler, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Atherton, California
  - Buena Park, California
  - Fresno, California
  - La Mesa, California
  - Los Angeles, California
  - Newport Beach, California
  - San Bernardino, California
  - San Diego, California
  - Tarzana, California
  - Torrance, California
  - Denver, Colorado
  - New Britain, Connecticut
  - Waterbury, Connecticut
  - Aventura, Florida
  - Clearwater, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Wellington, Florida
  - West Palm Beach, Florida
  - Alpharetta, Georgia
  - Roswell, Georgia
  - Melrose Park, Illinois
  - Fort Wayne, Indiana
  - Jeffersonville, Indiana
  - West Des Moines, Iowa
  - Overland Park, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Madisonville, Kentucky
  - Shreveport, Louisiana
  - Springfield, Massachusetts
  - Watertown, Massachusetts
  - Billings, Montana
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Lawrenceville, New Jersey
  - Albuquerque, New Mexico
  - Binghamton, New York
  - Garden City, New York
  - Kingston, New York
  - New York, New York
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Lyndhurst, Ohio
  - Wadsworth, Ohio
  - Bethany, Oklahoma
  - Edmond, Oklahoma
  - Bala-Cynwyd, Pennsylvania
  - Philadelphia, Pennsylvania
  - West Reading, Pennsylvania
  - Warwick, Rhode Island
  - Greer, South Carolina
  - Simpsonville, South Carolina
  - Arlington, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Virginia Beach, Virginia
  - Mountlake Terrace, Washington
  - Seattle, Washington
  - Spokane, Washington
- Canada (14):
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Bathurst, New Brunswick
  - Saint John, New Brunswick
  - Barrie, Ontario
  - Brampton, Ontario
  - Brantford, Ontario
  - Kitchener, Ontario
  - North Bay, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Granby, Quebec
  - Sherbrooke, Quebec
- Czechia (3):
  - Olomouc
  - Ostrava
  - Prague
- Denmark (4):
  - Aalborg
  - Aarhus N
  - Frederiksberg
  - Holstebro
- Finland (3):
  - Helsinki
  - Oulu
  - Tampere
- Germany (13):
  - Bad Ems
  - Eisleben Lutherstadt
  - Frankfurt
  - Hagenow
  - Halle
  - Henningsdorf
  - Hettstedt
  - Koblenz
  - Leipzig
  - Neunkirchen
  - Neustadt in Sachsen
  - Radebeul
  - Sangerhausen
- Hungary (8):
  - Budapest
  - Körmend
  - Nyíregyháza
  - Sopron
  - Szekszárd
  - Szentes
  - Székesfehérvár
  - Tatabánya
- Norway (3):
  - Bergen
  - Hamar
  - Tønsberg
- Slovakia (3):
  - Martin
  - Trenčín
  - Žilina
- Spain (6):
  - Barcelona
  - Coslada
  - Getafe Madrid
  - Gran Canaria
  - Madrid
  - Vic
- Sweden (6):
  - Gothenburg
  - Huddinge
  - Jönköping
  - Karlshamn
  - Malmo
  - Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Desroziers K, Aballea S, Maman K, Nazir J, Odeyemi I, Hakimi Z. Estimating EQ-5D and OAB-5D health state utilities for patients with overactive bladder. Health Qual Life Outcomes. 2013 Nov 19;11:200. doi: 10.1186/1477-7525-11-200. PMID 24246044
- [Derived] Herschorn S, Barkin J, Castro-Diaz D, Frankel JM, Espuna-Pons M, Gousse AE, Stolzel M, Martin N, Gunther A, Van Kerrebroeck P. A phase III, randomized, double-blind, parallel-group, placebo-controlled, multicentre study to assess the efficacy and safety of the beta(3) adrenoceptor agonist, mirabegron, in patients with symptoms of overactive bladder. Urology. 2013 Aug;82(2):313-20. doi: 10.1016/j.urology.2013.02.077. Epub 2013 Jun 13. PMID 23769122
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=26

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After screening, 2030 patients took placebo run-in study drug in a 2-week, single-blind, placebo run-in period. On completion of the run-in period, 1306 eligible patients were randomly assigned to receive placebo, mirabegron 25 mg or mirabegron 50 mg for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Started | 433 | 433 | 440
Safety Analysis Set (SAF) | 433 (All randomized patients who took at least 1 dose of double-blind study drug.) | 432 (All randomized patients who took at least 1 dose of double-blind study drug.) | 440 (All randomized patients who took at least 1 dose of double-blind study drug.)
Full Analysis Set (FAS) | 415 (Treated patients with a baseline and at least 1 post-baseline micturition measurement.) | 410 (Treated patients with a baseline and at least 1 post-baseline micturition measurement.) | 426 (Treated patients with a baseline and at least 1 post-baseline micturition measurement.)
Full Analysis Set Incontinence (FAS-I) | 262 (Full analysis set patients who had at least 1 incontinence episode at Baseline.) | 254 (Full analysis set patients who had at least 1 incontinence episode at Baseline.) | 257 (Full analysis set patients who had at least 1 incontinence episode at Baseline.)
Completed | 367 | 387 | 386
Not Completed | 66 | 46 | 54
Not completed — Eligibility criterion not met | 1 | 1 | 0
Not completed — Adverse Event | 15 | 18 | 12
Not completed — Lack of Efficacy | 11 | 4 | 3
Not completed — Withdrawal by Subject | 20 | 12 | 18
Not completed — Lost to Follow-up | 4 | 3 | 3
Not completed — Protocol Violation | 5 | 3 | 8
Not completed — Taking exclusionary medications | 7 | 4 | 8
Not completed — Medical History | 1 | 0 | 0
Not completed — Non-compliance with study procedures | 2 | 0 | 0
Not completed — Violation of exclusion criterion | 0 | 0 | 2
Not completed — Randomized but never received study drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Total
Number analyzed (Participants) | 433 | 432 | 440 | 1305
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline Measure data are provided for all randomized patients who took at least 1 dose of double-blind study drug (Safety Analysis Set).
  years | 58.2 (13.73) | 58.5 (12.85) | 60.3 (12.22) | 59.0 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 301 | 293 | 303 | 897
  Male | 132 | 139 | 137 | 408
Race/Ethnicity, Customized [Number; unit: participants]
  White | 389 | 394 | 400 | 1183
  Black or African American | 35 | 32 | 33 | 100
  Asian | 7 | 5 | 5 | 17
  Other | 2 | 1 | 2 | 5
Type of overactive bladder (OAB) [Number; unit: participants]
  Urge Incontinence | 126 | 168 | 169 | 463
  Mixed | 145 | 129 | 154 | 428
  Frequency | 162 | 135 | 117 | 414
Duration of OAB symptoms [Mean (Standard Deviation); unit: months] | 91.3 (96.82) | 96.3 (113.77) | 92.7 (97.88) | 93.4 (103.02)
Mean number of micturitions per 24 hours [Mean (Standard Deviation); unit: micturitions] — The average number of micturitions (urinations) recorded by the patient in a micturition diary for 3 days prior to the Baseline visit.
  micturitions | 11.54 (2.979) | 11.66 (3.117) | 11.69 (3.227) | 11.63 (3.108)
Mean volume voided per micturition [Mean (Standard Deviation); unit: mL] — Recorded by the patient in a micturition diary for 3 days prior to the Baseline visit.
  mL | 163.5 (56.39) | 165.4 (57.24) | 158.4 (52.17) | 162.4 (55.33)
Mean number of urgency episodes (grade 3 or 4) per 24 hours [Mean (Standard Deviation); unit: urgency episodes] — Urgency episodes were those classified by the patient in a 3-day micturition diary as 3 or 4 on the Patient Perception of Intensity of Urgency (PPIUS) scale: 0: No urgency; 1: Mild urgency; 2: Moderate urgency, could delay voiding a short while; 3: Severe urgency, could not delay voiding; 4: Urge incontinence, leaked before arriving to the toilet.
  urgency episodes | 5.43 (3.335) | 5.54 (3.622) | 5.81 (3.559) | 5.60 (3.508)
Mean level of urgency [Mean (Standard Deviation); unit: scores on a scale] — Average of patients' ratings on the degree of associated urgency for each micturition and/or incontinence episode recorded in a 3-day micturition diary according to the following 5-point categorical scale (Patient Perception of Intensity of Urgency Scale): 0: No urgency; 1: Mild urgency; 2: Moderate urgency, could delay voiding a short while; 3: Severe urgency, could not delay voiding; 4: Urge incontinence, leaked before arriving to the toilet.
  scores on a scale | 2.36 (0.550) | 2.37 (0.573) | 2.41 (0.556) | 2.38 (0.560)
Mean number of nocturia episodes per 24 hours [Mean (Standard Deviation); unit: nocturia episodes] — The average number of times a patient woke at night to urinate (excluding incontinence only episodes) recorded for 3 days prior to the Baseline visit in the patient micturition diary.
  nocturia episodes | 1.82 (1.332) | 1.94 (1.552) | 2.03 (1.528) | 1.93 (1.465)
Mean number of pads used per 24 hours [Mean (Standard Deviation); unit: pads] — Recorded by the patient in a micturition diary for 3 days prior to the Baseline visit.
  pads | 0.91 (1.786) | 0.79 (1.449) | 0.84 (1.700) | 0.85 (1.666)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment (Final Visit) in Mean Number of Incontinence Episodes Per 24 Hours
Description: The average number of incontinence episodes (any involuntary leakage of urine) per day was derived from the number of incontinence episodes recorded by the patient in a micturition diary for 3-days before the Baseline and Week 12 clinic visits. Least Squares (LS) Means were generated from an analysis of covariance (ANCOVA) model with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Week 12
Population: The full analysis set-Incontinence included all randomized patients who took at least 1 dose of double-blind study drug and who had a baseline and at least 1 post baseline micturition measurement in the visit diary and who had at least 1 incontinence episode at baseline. Last observation carried forward (LOCF) was utilized.
Measure: Least Squares Mean (Standard Error); unit: Incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 262 | 254 | 257
Incontinence episodes | -0.96 (0.122) | -1.36 (0.124) | -1.38 (0.123)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 25 mg; Since there were 2 coprimary efficacy endpoints and 6 key secondary efficacy endpoints, the multiplicity among the endpoints was controlled at a type I error rate at the alpha = 0.05 level using a stepwise parallel gatekeeping procedure (8 stages). In addition, since two mirabegron treatment groups were compared with placebo per endpoint, the Hochberg procedure was used to adjust for multiplicity. A stratified rank ANCOVA model was utilized for hypothesis testing; Test type: Superiority or Other; p = 0.005, Stratified rank ANCOVA — The response variable for the stratified rank ANCOVA was standardized ranks on change from Baseline to Final Visit value with baseline standardized ranks and gender as covariates and geographic region as a stratum; LS mean difference was derived from an ANCOVA model with treatment group, gender, and geographic region as fixed factors and baseline as a covariate; LS Mean Difference = -0.40, 95% CI 2-sided [-0.74 to -0.06]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 50 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, Stratified rank ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.42, 95% CI 2-sided [-0.76 to -0.08]

2. Secondary Outcome: Change From Baseline to End of Treatment (Final Visit) in Mean Volume Voided Per Micturition
Description: The average volume voided per micturition was calculated from the volume of each micturition measured by the patient and recorded in a micturition diary for 3 days before the Baseline and Week 12 clinic visits. LS Means were generated from an ANCOVA model with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Week 12
Population: The full analysis set included all randomized patients who took at least 1 dose of double-blind study drug and who had a baseline and at least 1 post baseline micturition measurement in the visit diary. Last observation carried forward was utilized.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
mL | 8.3 (2.23) | 12.8 (2.24) | 20.7 (2.20)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 25 mg; Since there were 2 coprimary efficacy endpoints and 6 key secondary efficacy endpoints, the multiplicity among the endpoints was controlled at a type I error rate at the alpha = 0.05 level using a stepwise parallel gatekeeping procedure (8 stages). In addition, since two mirabegron treatment groups were compared with placebo per endpoint, the Hochberg procedure was used to adjust for multiplicity. An ANCOVA model was used for hypothesis testing; Test type: Superiority or Other; p = 0.15, ANCOVA — LS mean difference and p-value were derived from an ANCOVA model with treatment group, gender, and geographic region as fixed factors and baseline as a covariate; LS Mean Difference = 4.6, 95% CI 2-sided [-1.6 to 10.8]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 12.4, 95% CI 2-sided [6.3 to 18.6]

3. Primary Outcome: Change From Baseline to End of Treatment (Final Visit) in Mean Number of Micturitions Per 24 Hours
Description: The average number of micturitions (urinations) per 24 hours was derived from the number of times a patient urinates (excluding incontinence only episodes) per day recorded by the patient in a micturition diary for 3-days before the Baseline and Week 12 clinic visits. LS Means generated from an ANCOVA model with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
micturitions | -1.18 (0.124) | -1.65 (0.125) | -1.60 (0.122)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 25 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.007, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.47, 95% CI 2-sided [-0.82 to -0.13]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.42, 95% CI 2-sided [-0.76 to -0.08]

4. Secondary Outcome: Change From Baseline to Week 4 in Mean Number of Incontinence Episodes Per 24 Hours
Description: The average number of incontinence episodes (any involuntary leakage of urine) per 24 hours was derived from the number of incontinence episodes recorded by the patient in a micturition diary for 3-days before the Baseline and Week 4 clinic visits. LS Means were generated from an ANCOVA model with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Week 4
Population: The full analysis set-Incontinence included all randomized patients who took at least 1 dose of double-blind study drug and who had a baseline and at least 1 post baseline micturition measurement in the visit diary and who had at least 1 incontinence episode at baseline. Last observation carried forward (LOCF) was not utilized in this analysis.
Measure: Least Squares Mean (Standard Error); unit: Incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 262 | 254 | 255
Incontinence episodes | -0.62 (0.120) | -0.96 (0.122) | -1.13 (0.122)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.039, Stratified rank ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.34, 95% CI 2-sided [-0.68 to -0.01]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 50 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Stratified rank ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.51, 95% CI 2-sided [-0.85 to -0.17]

5. Secondary Outcome: Change From Baseline to Week 4 in Mean Number of Micturitions Per 24 Hours
Description: The average number of micturitions (urinations) per 24 hours was calculated from the number of micturitions recorded by the patient in a micturition diary for 3-days before the Baseline and Week 4 clinic visits. LS Means generated from an ANCOVA model with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Week 4
Population: The full analysis set included all randomized patients who took at least 1 dose of double-blind study drug and who had a baseline and at least 1 post baseline micturition measurement in the visit diary. Last observation carried forward was not utilized in this analysis.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 424
micturitions | -0.78 (0.124) | -0.96 (0.124) | -1.14 (0.122)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 25 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.30, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Difference = -0.18, 95% CI 2-sided [-0.53 to 0.16]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.035, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean Difference = -0.37, 95% CI 2-sided [-0.71 to -0.03]

6. Secondary Outcome: Change From Baseline to End of Treatment (Final Visit) in Mean Level of Urgency
Description: Average of patients' ratings on the degree of urgency associated with each micturition and/or incontinence episode recorded in a 3-day micturition diary according to the following 5-point categorical scale (Patient Perception of Intensity of Urgency Scale): 0: No urgency; 1: Mild urgency; 2: Moderate urgency, could delay voiding a short while; 3: Severe urgency, could not delay voiding; 4: Urge incontinence, leaked before arriving to the toilet. LS Means are from an ANCOVA with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 413 | 410 | 426
scores on a scale | -0.15 (0.028) | -0.22 (0.029) | -0.29 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 25 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.083, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean Difference = -0.07, 95% CI 2-sided [-0.15 to 0.01]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.14, 95% CI 2-sided [-0.22 to -0.06]

7. Secondary Outcome: Change From Baseline to End of Treatment (Final Visit) in Mean Number of Urgency Incontinence Episodes Per 24 Hours
Description: The involuntary leakage of urine accompanied by or immediately proceeded by urgency, derived from the number of incontinence episodes classified by the patient in a 3-day micturition diary as 3 or 4 on the Patient Perception of Intensity of Urgency Scale: 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could postpone voiding a short while; 3 = Severe urgency, could not postpone voiding; 4 = Urge incontinence, leaked before arriving to the toilet. LS Means are from an ANCOVA with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Week 12
Population: The full analysis set-Incontinence included all randomized patients who took at least 1 dose of double-blind study drug and who had a baseline and at least 1 post baseline micturition measurement in the visit diary and who had at least 1 urgency incontinence episode at baseline. Last observation carried forward (LOCF) was utilized.
Measure: Least Squares Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 256 | 247 | 251
urgency incontinence episodes | -0.95 (0.110) | -1.31 (0.112) | -1.33 (0.111)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, Stratified rank ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.36, 95% CI 2-sided [-0.67 to -0.05]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 50 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Stratified rank ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.39, 95% CI 2-sided [-0.69 to -0.08]

8. Secondary Outcome: Change From Baseline to End of Treatment (Final Visit) in Mean Number of Urgency Episodes (Grades 3 or 4) Per 24 Hours
Description: The average number of urgency episodes (the sudden, compelling desire to pass urine, which is difficult to defer), derived from urgency episodes classified by the patient in a 3-day micturition diary as grade 3 or 4 on the Patient Perception of Intensity of Urgency Scale: 0: No urgency; 1: Mild urgency; 2: Moderate urgency, could delay voiding a short while; 3: Severe urgency, could not delay voiding; 4: Urge incontinence, leaked before arriving to the toilet. LS Means are from an ANCOVA with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Week 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 post baseline micturition measurement in the visit diary and at least 1 episode of urgency grade 3 or 4 at baseline. Last observation carried forward was utilized.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 413 | 410 | 426
urgency episodes | -1.35 (0.154) | -1.68 (0.155) | -1.94 (0.152)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 25 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.13, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.33, 95% CI 2-sided [-0.76 to 0.10]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.007, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.59, 95% CI 2-sided [-1.01 to -0.16]

9. Secondary Outcome: Change From Baseline to Week 8 and Week 12 in Mean Number of Micturitions Per 24 Hours
Description: The average number of micturitions (urinations) per 24 hours was calculated from the number of micturitions recorded by the patient in a micturition diary for 3-days before the Baseline, Week 8 and 12 clinic visits. LS Means were generated from an ANCOVA model with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Weeks 8 and 12
Population: The full analysis set included all randomized patients who took at least 1 dose of double-blind study drug and who had a baseline and at least 1 post baseline micturition measurement in the visit diary. The number of patients included in the calculation for each time point is noted as "N". LOCF was not used in this analysis.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
micturitions
  Week 8 [N= 377; 395; 399] | -1.09 (0.130) | -1.52 (0.127) | -1.53 (0.127)
  Week 12 [N= 366; 387; 386] | -1.47 (0.122) | -1.68 (0.119) | -1.69 (0.119)

10. Secondary Outcome: Change From Baseline to Week 8 and Week 12 in Mean Number of Incontinence Episodes Per 24 Hours
Description: The average number of incontinence episodes (any involuntary leakage of urine) per 24 hours was derived from the number of incontinence episodes recorded by the patient in a micturition diary for 3-days before the Baseline, Week 8 and Week 12 clinic visits. LS Means were generated from an ANCOVA model with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Weeks 8 and 12
Population: The full analysis set-incontinence included all randomized patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 post baseline micturition measurement in the visit diary and at least 1 incontinence episode at baseline. The number of patients included at each time point is noted as "N". LOCF was not utilized.
Measure: Least Squares Mean (Standard Error); unit: Incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 262 | 254 | 257
Incontinence episodes
  Week 8 [N= 236; 244; 241] | -1.04 (0.117) | -1.38 (0.116) | -1.39 (0.116)
  Week 12 [N= 231; 239; 232] | -1.08 (0.120) | -1.36 (0.118) | -1.43 (0.119)

11. Secondary Outcome: Change From Baseline to Week 4, Week 8 and Week 12 in Mean Volume Voided Per Micturition
Description: The average volume voided per micturition was calculated from the volume of each micturition measured by the patient and recorded in a micturition diary for 3 days before the Baseline and Week 4, 8 and 12 clinic visits. LS Means generated from an ANCOVA model with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The full analysis set included all randomized patients who took at least 1 dose of double-blind study drug and who had a baseline and at least 1 post baseline micturition measurement in the visit diary. LOCF was not utilized in this analysis. The number of participants included in the calculation for each time point is noted as "N".
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
mL
  Week 4 [N=415; 410; 424] | 7.6 (1.85) | 10.6 (1.86) | 17.8 (1.83)
  Week 8 [N=377; 395; 399] | 9.8 (2.21) | 15.7 (2.16) | 17.9 (2.15)
  Week 12 [N=366; 387; 386] | 8.2 (2.41) | 13.6 (2.34) | 22.5 (2.34)

12. Secondary Outcome: Change From Baseline to Week 4, Week 8 and Week 12 in Mean Number of Urgency Incontinence Episodes Per 24 Hours
Description: as for outcome 7
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The full analysis set-Incontinence included all randomized patients who took at least 1 dose of double-blind study drug and who had a baseline and at least 1 post baseline micturition measurement in the visit diary and who had at least 1 urgency incontinence episode (grade 3 or 4) at baseline. LOCF was not utilized.
Measure: Least Squares Mean (Standard Error); unit: Urgency incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 262 | 254 | 257
Urgency incontinence episodes
  Week 4 [N=256; 247; 249] | -0.63 (0.107) | -0.98 (0.109) | -1.12 (0.109)
  Week 8 [N=231; 237; 236] | -1.02 (0.101) | -1.33 (0.100) | -1.39 (0.100)
  Week 12 [N=226; 232; 227] | -1.06 (0.105) | -1.32 (0.104) | -1.39 (0.104)

13. Secondary Outcome: Change From Baseline to Week 4, Week 8 and Week 12 in Mean Number of Urgency Episodes (Grades 3 or 4) Per 24 Hours
Description: as for outcome 8
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 post baseline micturition measurement in the visit diary and at least 1 episode of urgency grade 3 or 4 at baseline. LOCF was not utilized for this analysis. N is the number of patients included at each time point.
Measure: Least Squares Mean (Standard Error); unit: Urgency episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
Urgency episodes
  Week 4 [N=412; 409; 423] | -0.90 (0.143) | -0.97 (0.143) | -1.47 (0.141)
  Week 8 [N=377; 393; 398] | -1.17 (0.162) | -1.51 (0.159) | -1.73 (0.158)
  Week 12 [N=364; 385; 385] | -1.60 (0.162) | -1.72 (0.157) | -1.99 (0.157)

14. Secondary Outcome: Change From Baseline to Week 4, Week 8 and Week 12 in Mean Level of Urgency
Description: as for outcome 6
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The full analysis set included all randomized patients who took at least 1 dose of double-blind study drug and who had a baseline and at least 1 post baseline micturition measurement in the visit diary. LOCF was not utilized for this analysis. The number of participants included in the calculation for each time point is noted as "N".
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
scores on a scale
  Week 4 [N=412; 409; 423] | -0.10 (0.025) | -0.12 (0.025) | -0.20 (0.025)
  Week 8 [N=377; 393; 398] | -0.15 (0.029) | -0.19 (0.028) | -0.26 (0.028)
  Week 12 [N=364; 385; 385] | -0.19 (0.030) | -0.23 (0.029) | -0.30 (0.029)

15. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and Final Visit in Mean Number of Nocturia Episodes Per 24 Hours
Description: Nocturia is defined as waking at night one or more times to void. The average number of times a patient urinated (excluding incontinence only episodes) during sleeping time per day was derived from the 3-day patient micturition diary.
  LS Means are from an ANCOVA with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 post baseline micturition measurement in the visit diary and who had at least one nocturia episode at baseline. LOCF was used for the Final Visit analysis. N is the number of participants included at each time point.
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
nocturia episodes
  Week 4 [N=362; 362; 376] | -0.30 (0.059) | -0.27 (0.058) | 0.38 (0.057)
  Week 8 [N=329; 349; 354] | -0.45 (0.059) | -0.41 (0.057) | -0.44 (0.057)
  Week 12 [N=321; 342; 344] | -0.54 (0.058) | -0.50 (0.056) | -0.52 (0.056)
  Final Visit (LOCF) [N=362; 362; 378] | -0.48 (0.058) | -0.49 (0.058) | -0.52 (0.057)

16. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and Final Visit in Mean Number of Pads Used Per 24 Hours
Description: The average number of times a patient records a new pad used per day during the 3-day micturition diary period.
  LS Means are from an ANCOVA with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 postbaseline micturition measurement in the visit diary and who had at least one use of a pad at baseline. LOCF was used for the Final Visit analysis. N is the number of participants included at each time point.
Measure: Least Squares Mean (Standard Error); unit: pads
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
pads
  Week 4 [N=145; 136; 136] | -0.72 (0.117) | -0.59 (0.121) | -0.81 (0.120)
  Week 8 [N=131; 131; 128] | -0.97 (0.119) | -0.79 (0.119) | -1.16 (0.120)
  Week 12 [N=129; 129; 124] | -1.06 (0.125) | -0.89 (0.125) | -1.17 (0.127)
  Final Visit (LOCF) [N=145; 136; 137] | -0.99 (0.118) | -0.83 (0.122) | -1.16 (0.121)

17. Secondary Outcome: Percentage of Participants With Zero Incontinence Episodes at Weeks 4, 8, 12 and the Final Visit
Description: The percentage of participants with no incontinence episodes for the 3 days prior to each clinic visit derived from the micturition diary recorded by the patient.
Time Frame: Weeks 4, 8 and 12
Population: The full analysis set-incontinence included all patients who took at least 1 dose of double-blind study drug & had a baseline & at least 1 postbaseline micturition measurement in the visit diary & who had at least 1 incontinence episode at baseline. LOCF was used for the Final Visit analysis. N is the number of patients included at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 262 | 254 | 257
percentage of participants
  Week 4 [N=262; 254; 255] | 28.2 | 31.5 | 36.5
  Week 8 [N=236; 244; 241] | 41.9 | 44.7 | 41.9
  Week 12 [N=231; 239; 232] | 42.0 | 46.9 | 47.4
  Final Visit (LOCF) [N=262; 254; 257] | 39.7 | 45.7 | 47.1

18. Secondary Outcome: Percentage of Participants With ≥ 50% Reduction in Incontinence Episodes at Weeks 4, 8, 12 and the Final Visit
Description: The percentage of participants with at least a 50% decrease from baseline in mean number of incontinence episodes per 24 hours during the 3 days prior to each clinic visit derived from the patient micturition diary.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 262 | 254 | 255
percentage of participants
  Week 4 [N=262; 254; 255] | 46.6 | 54.7 | 61.6
  Week 8 [N=236; 244; 241] | 62.7 | 71.7 | 71.4
  Week 12 [N=231; 239; 232] | 61.5 | 74.1 | 71.1
  Final Visit (LOCF) [N=262; 254; 257] | 59.2 | 72.8 | 70.0

19. Secondary Outcome: Percentage of Responders for Mean Level of Urgency
Description: Percentage of participants with a decrease from Baseline to Final Visit in mean level of urgency at least as large as the pre-specified minimally important difference (MID). The MID was determined to be 0.24 for mean level of urgency. Mean level of urgency was derived from the average of patients' ratings on the degree of urgency associated with each micturition and/or incontinence episode recorded in a 3-day micturition diary according to the Patient Perception of Intensity of Urgency Scale which ranged from 0 (No urgency) to 4 (Urge incontinence).
Time Frame: Baseline and Week 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug & had a baseline & at least 1 postbaseline micturition measurement in the visit diary. LOCF was used for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 413 | 410 | 426
percentage of participants | 36.6 | 40.5 | 44.8

20. Secondary Outcome: Percentage of Responders for Number of Grade 3 or 4 Urgency Episodes
Description: Percentage of participants with a decrease from baseline to final visit in mean number of urgency episodes (grade 3 or 4) at least as large as the pre-specified minimally important difference (MID). The MID was determined to be 1.54 for mean number of urgency episodes (grade 3 or 4). The mean number of urgency episodes was derived from urgency episodes classified by the patient in a 3-day micturition diary as grade 3 or 4 on the Patient Perception of Intensity of Urgency Scale where a score 3=severe urgency and 4=urge incontinence.
Time Frame: Baseline and Week 12
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 413 | 410 | 426
percentage of participants | 44.6 | 47.1 | 57.7

21. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and Final Visit in Symptom Bother Score
Description: Overactive bladder symptoms were assessed using the symptom bother scale of the overactive bladder questionnaire. The symptom bother scale consists of 8 questions answered by the participant on a scale from 1-6. The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 to 100, with 100 indicating worst severity. A negative change from Baseline in symptom bother score indicates improvements.
  LS Means are from an ANCOVA with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 postbaseline micturition measurement in the visit diary. LOCF was used for the Final Visit analysis. The number of participants included in the calculation for each time point is noted as "N".
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
scores on a scale
  Week 4 [N=402; 406; 418] | -12.2 (0.82) | -13.7 (0.82) | -12.7 (0.80)
  Week 8 [N=376; 389; 391] | -15.1 (0.92) | -17.4 (0.91) | -18.5 (0.90)
  Week 12 [N=360; 380; 378] | -17.5 (0.94) | -18.0 (0.91) | -19.6 (0.92)
  Final Visit (LOCF) [N=405; 407; 422] | -16.0 (0.90) | -17.9 (0.90) | -18.8 (0.88)

22. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and Final Visit in Health-related Quality of Life (HRQL) Total Score
Description: Health-related quality of life was assessed by the HRQL subscales (coping, concern, sleep and social interaction) of the overactive bladder questionnaire (OABq). The HRQL total score was calculated by adding the 4 HRQL subscale scores, and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from Baseline in HRQL score indicates improvements.
  LS Means are from an ANCOVA with treatment group, gender, and geographic region as fixed factors and baseline as a covariate.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
scores on a scale
  Week 4 [N=403; 408; 417] | 8.8 (0.73) | 11.4 (0.73) | 9.2 (0.72)
  Week 8 [N=373; 393; 390] | 12.1 (0.82) | 14.3 (0.80) | 13.8 (0.80)
  Week 12 [N=360; 383; 377] | 13.8 (0.84) | 14.4 (0.81) | 14.7 (0.82)
  Final Visit (LOCF) [N=406; 408; 419] | 13.0 (0.80) | 14.3 (0.79) | 14.2 (0.78)

23. Secondary Outcome: Change From Baseline to Week 12 and Final Visit in Work Productivity and Activity Impairment (WPAI): Percent Work Time Missed
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess the degree and extent to which overactive bladder (OAB) symptoms interfered with work productivity in the last 7 days. Percent of work time missed is derived from the number of hours of work missed due to OAB symptoms as a percentage of total hours that should have been worked. A higher percentage indicates more hours missed. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug & had a baseline & at least 1 postbaseline micturition measurement in the visit diary. The number of patients at each time point (N) includes those with both baseline and post-baseline values who were employed. LOCF was used for the Final Visit analysis.
Measure: Mean (Standard Deviation); unit: percent work time missed
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
percent work time missed
  Week 12 [N=112; 118; 118] | 0.6 (14.42) | 0.7 (15.63) | -1.5 (7.45)
  Final Visit (LOCF) [N=119; 122; 123] | 0.6 (14.01) | 0.7 (15.37) | -1.3 (7.35)

24. Secondary Outcome: Change From Baseline to Week 12 and Final Visit in Work Productivity and Activity Impairment (WPAI): Percent Impairment While Working
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess the degree and extent to which overactive bladder (OAB) symptoms interfered with work productivity in the last 7 days. Percent impairment while working was derived from the patient's assessment of the degree to which OAB affected their productivity while working. A higher percentage indicates greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent impairment while working
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
percent impairment while working
  Week 12 [N=123; 130; 128] | -11.6 (26.44) | -10.2 (22.01) | -13.0 (23.89)
  Final Visit (LOCF) [N=130; 135; 134] | -11.5 (26.09) | -10.1 (21.67) | -13.1 (23.60)

25. Secondary Outcome: Change From Baseline to Week 12 and Final Visit in Work Productivity and Activity Impairment (WPAI): Percent Overall Work Impairment
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess the degree and extent to which overactive bladder (OAB) symptoms interfered with work productivity in the last 7 days. Percent overall work impairment takes into account both hours missed due to OAB symptoms and the patient's assessment of the degree to which OAB affected their productivity while working. A higher percentage indicates greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent overall work impairment
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
percent overall work impairment
  Week 12 [N=110; 115; 118] | -14.1 (26.57) | -11.0 (23.65) | -13.3 (24.45)
  Final Visit (LOCF) [N=117; 119; 123] | -13.8 (26.18) | -10.8 (23.33) | -13.3 (24.21)

26. Secondary Outcome: Change From Baseline to Week 12 and Final Visit in Work Productivity and Activity Impairment (WPAI): Percent Activity Impairment
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess the degree and extent to which overactive bladder (OAB) symptoms interfered with daily activities over the last 7 days. Percent activity impairment is derived from the patient's assessment of the degree to which OAB affected their regular daily activities. A higher percentage indicates greater impairment. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 postbaseline micturition measurement in the visit diary. The number of participants at each time point (N) included patients with both baseline and post-baseline values. LOCF was used for the Final Visit analysis.
Measure: Mean (Standard Deviation); unit: percent activity impairment
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
percent activity impairment
  Week 12 [N=353; 366; 362] | -11.4 (26.66) | -12.3 (26.10) | -13.1 (26.22)
  Final Visit (LOCF) [N=373; 376; 378] | -11.0 (26.87) | -11.9 (26.18) | -13.3 (26.12)

27. Secondary Outcome: Change From Baseline to Final Visit in European Quality of Life-5 Dimensions (EQ-5D) Mobility Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state:
  I have no problems in walking about; I have some problems in walking about; I am confined to bed.
  In the table below, each row title lists Baseline health status first followed by Final Visit health status and reports the number of patients in that category. Missing data indicates patients with no data available for that Visit.
Time Frame: Baseline and Week 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 postbaseline micturition measurement in the visit diary. LOCF was used for this analysis.
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
participants
  No problem -> No problem | 327 | 310 | 304
  No problem -> Some problems | 16 | 20 | 33
  No problem -> Confined to bed | 0 | 0 | 0
  No problem -> Missing data | 6 | 1 | 2
  Some problems -> No problems | 22 | 31 | 36
  Some problems -> Some problems | 39 | 45 | 48
  Some problems -> Confined to bed | 0 | 0 | 1
  Some problems -> Missing data | 1 | 0 | 2
  Confined -> No problems | 1 | 0 | 0
  Confined -> Some problems | 0 | 0 | 0
  Confined -> Confined to bed | 0 | 0 | 0
  Confined -> Missing data | 0 | 0 | 0
  Missing data -> No problem | 3 | 3 | 0
  Missing data -> Some problems | 0 | 0 | 0
  Missing data -> Confined to bed | 0 | 0 | 0
  Missing data -> Missing data | 0 | 0 | 0

28. Secondary Outcome: Change From Baseline to Final Visit in European Quality of Life-5 Dimensions (EQ-5D) Self-Care Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state:
  I have no problems with self-care; I have some problems washing or dressing myself; I am unable to wash or dress myself. In the table below, each row title lists Baseline health status first followed by Final Visit health status and reports the number of patients in that category. Missing data indicates patients with no data available for that Visit.
Time Frame: Baseline and Week 12
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
participants
  No problem -> No problem | 389 | 385 | 403
  No problem -> Some problems | 5 | 10 | 6
  No problem -> Unable to wash or dress myself | 0 | 0 | 1
  No problem -> Missing data | 7 | 1 | 4
  Some problems -> No problems | 5 | 3 | 2
  Some problems -> Some problems | 6 | 8 | 9
  Some problems -> Unable to wash or dress myself | 0 | 0 | 0
  Some problems -> Missing data | 0 | 0 | 0
  Unable to wash or dress myself -> No problems | 0 | 0 | 0
  Unable to wash or dress myself -> Some problems | 0 | 0 | 1
  Unable to wash or dress -> Unable to wash or dress | 0 | 0 | 0
  Unable to wash or dress myself -> Missing data | 0 | 0 | 0
  Missing data -> No problem | 3 | 3 | 0
  Missing data -> Some problems | 0 | 0 | 0
  Missing data -> Unable to wash or dress myself | 0 | 0 | 0
  Missing data -> Missing data | 0 | 0 | 0

29. Secondary Outcome: Change From Baseline to Final Visit in European Quality of Life-5 Dimensions (EQ-5D) Usual Activities Score
Description: The EQ-5D is a standardized, nondisease-specific instrument for describing health status. Participants were asked which statement best describes their health state with regard to usual activities (work, study or leisure): I have no problems performing my usual activities; I have some problems performing my usual activities; I am unable to perform my usual activities. In the table below, each row title lists Baseline health status first followed by Final Visit health status and reports the number of patients in that category. Missing data indicates patients with no data available at that Visit.
Time Frame: Baseline and Week 12
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
participants
  No problem -> No problem | 313 | 303 | 293
  No problem -> Some problems | 27 | 27 | 31
  No problem -> Unable to perform usual activities | 0 | 1 | 0
  No problem -> Missing data | 6 | 0 | 4
  Some problems -> No problems | 35 | 38 | 51
  Some problems -> Some problems | 30 | 35 | 44
  Some problems->Unable to perform usual activities | 0 | 1 | 1
  Some problems -> Missing data | 1 | 0 | 0
  Unable to perform usual activities -> No problems | 0 | 0 | 0
  Unable to perform usual activities-> Some problems | 0 | 1 | 1
  Unable to perform -> Unable to perform | 0 | 0 | 1
  Unable to perform usual activities -> Missing data | 0 | 1 | 0
  Missing data -> No problem | 3 | 2 | 0
  Missing data -> Some problems | 0 | 1 | 0
  Missing data -> Unable to perform usual activities | 0 | 0 | 0
  Missing data -> Missing data | 0 | 0 | 0

30. Secondary Outcome: Change From Baseline to Final Visit in European Quality of Life-5 Dimensions (EQ-5D) Pain/Discomfort Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state:
  I have no pain or discomfort; I have moderate pain or discomfort; I have extreme pain or discomfort. In the table below, each row title lists Baseline health status first followed by Final Visit health status and reports the number of patients in that category. Missing data indicates patients with no data available for that Visit.
Time Frame: Baseline and Week 12
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
participants
  No pain -> No pain | 209 | 200 | 185
  No pain -> Moderate pain | 34 | 36 | 41
  No pain -> Extreme pain | 2 | 4 | 3
  No pain -> Missing data | 4 | 0 | 3
  Moderate pain -> No pain | 58 | 65 | 75
  Moderate pain -> Moderate pain | 85 | 92 | 87
  Moderate pain -> Extreme pain | 5 | 0 | 7
  Moderate pain ->Missing data | 3 | 0 | 0
  Extreme pain -> No pain | 0 | 0 | 5
  Extreme pain -> Moderate pain | 9 | 4 | 13
  Extreme pain -> Extreme pain | 2 | 5 | 5
  Extreme pain -> Missing data | 0 | 1 | 1
  Missing data-> No pain | 2 | 1 | 1
  Missing data -> Moderate pain | 2 | 2 | 0
  Missing data -> Extreme pain | 0 | 0 | 0
  Missing data -> Missing data | 0 | 0 | 0

31. Secondary Outcome: Change From Baseline to Final Visit in European Quality of Life-5 Dimensions (EQ-5D) Anxiety/Depression Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state:
  I am not anxious or depressed; I am moderately anxious or depressed; I am extremely anxious or depressed. In the table below, each row title lists Baseline health status first followed by Final Visit health status and reports the number of patients in that category. Missing data indicates patients with no data available for that Visit.
Time Frame: Baseline and Week 12
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
participants
  Not anxious -> Not anxious | 239 | 243 | 225
  Not anxious -> Moderately anxious | 20 | 29 | 33
  Not anxious -> Extremely anxious | 1 | 1 | 3
  Not anxious -> Missing data | 3 | 0 | 4
  Moderately anxious -> Not anxious | 52 | 50 | 58
  Moderately anxious -> Moderately anxious | 77 | 74 | 89
  Moderately anxious -> Extremely anxious | 4 | 2 | 3
  Moderately anxious -> Missing data | 4 | 0 | 0
  Extremely anxious -> Not anxious | 1 | 1 | 2
  Extremely anxious -> Moderately anxious | 6 | 5 | 6
  Extremely anxious -> Extremely anxious | 4 | 1 | 3
  Extremely anxious -> Missing data | 0 | 1 | 0
  Missing data -> Not anxious | 3 | 2 | 0
  Missing data -> Moderately anxious | 1 | 1 | 0
  Missing data -> Extremely anxious | 0 | 0 | 0
  Missing data -> Missing data | 0 | 0 | 0

32. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and Final Visit in the European Quality of Life-5 Dimensions (EQ-5D) Visual Analog Scale (VAS)
Description: The EQ-5D is an international, standardized, generic instrument for describing and evaluating health status. Health status is assessed by patients evaluating their health on a vertical, visual analog scale from 0 to 100 where the endpoints are labeled 'Worst imaginable health state' (=0) and 'Best imaginable health state' (=100). On the EQ-5D VAS, a positive change from baseline indicates improvement.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug & had a baseline & at least 1 postbaseline micturition measurement in the visit diary. The number of participants at each time point (N) includes only patients with both baseline and post-baseline values. LOCF was used for the Final Visit analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
scores on a scale
  Week 4 [N=399; 401; 411] | 0.38 (15.312) | 2.43 (13.929) | 1.67 (13.712)
  Week 8 [N=368; 386; 383] | 3.14 (15.389) | 3.95 (15.766) | 4.13 (14.795)
  Week 12 [N=359; 379; 375] | 4.26 (15.535) | 4.40 (15.282) | 5.59 (17.112)
  Final Visit (LOCF) [N=404; 406; 419] | 3.43 (16.076) | 4.12 (15.082) | 4.96 (17.225)

33. Secondary Outcome: Change From Baseline to Week 12 and Final Visit in Patient Perception of Bladder Condition (PPBC)
Description: The PPBC scale is a global assessment tool that asks patients to rate their impression of their current bladder condition on a 6-point scale from 1: 'Does not cause me any problems at all'; 2: 'Causes me some very minor problems'; 3: 'Causes me some minor problems'; 4: 'Causes me (some) moderate problems'; 5: 'Causes me severe problems' and 6: 'Causes me many severe problems'. LS means are from an ANCOVA model with treatment group, gender, and geographical regions as fixed factors and baseline as a covariate. A negative change from Baseline score indicates improvement.
Time Frame: Baseline and Week 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 postbaseline micturition measurement in the visit diary. The number of participants included at each time point (N) only includes those with baseline and post-baseline values. LOCF was used for the Final Visit analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
scores on a scale
  Week 12 [N=357; 381; 378] | -0.7 (0.06) | -0.8 (0.06) | -0.8 (0.06)
  Final Visit (LOCF) [N=376; 391; 395] | -0.7 (0.06) | -0.8 (0.06) | -0.7 (0.06)

34. Secondary Outcome: Change From Baseline to Week 12 and Final Visit in Treatment Satisfaction on Visual Analog Scale (TS-VAS)
Description: The TS-VAS is a visual analog scale (VAS) that asks patients to rate their satisfaction with treatment by placing a vertical mark on a 10 cm line where the endpoints are labeled 'No, not at all' on the left (=0) to 'Yes, completely satisfied' on the right (=10). LS means are from an ANCOVA model with treatment group, gender, and geographical regions as fixed factors and baseline as a covariate. A positive change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
scores on a scale
  Week 12 [N=357; 379; 371] | 1.18 (0.156) | 1.58 (0.151) | 1.94 (0.153)
  Final Visit (LOCF) [N=377; 389; 388] | 1.05 (0.154) | 1.54 (0.152) | 1.88 (0.152)

35. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and Final Visit in Number of Non-study Related Visits to Physician
Description: The number of times the patient visited a physician's office during the 4 weeks prior to each study visit (excluding study visits) because of the patient's bladder condition.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 postbaseline micturition measurement in the visit diary. The number of participants at each time point (N) includes only patients with both baseline and post-baseline values. LOCF was used for the Final Visit analysis.
Measure: Mean (Standard Deviation); unit: Physician visits
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
Physician visits
  Week 4 [N=410; 410; 424] | 0.0 (0.30) | -0.0 (0.12) | -0.0 (0.16)
  Week 8 [N=381; 394; 399] | -0.0 (0.18) | -0.0 (0.13) | 0.0 (0.16)
  Week 12 [N=364; 386; 382] | -0.0 (0.17) | 0.0 (0.14) | -0.0 (0.13)
  Final Visit (LOCF) [N=410; 410; 424] | -0.0 (0.18) | 0.0 (0.15) | -0.0 (0.12)

36. Secondary Outcome: Summary of Baseline, Week 12 and Final Visit Change in Bladder Symptoms on the Clinician Global Impression Scale
Description: The Clinician Global Impression Scale (CGI) assessed the change in the patient's bladder symptoms since the start of the study and was completed by the physician at Baseline and at Week 12/end of treatment. The degree of change was categorized as one of the following: 'Very much improved', 'Much improved', 'Minimally improved', 'No change', 'Minimally worse', 'Much worse', or 'Very much worse'.
Time Frame: Baseline and Week 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 postbaseline micturition measurement in the visit diary. This assessment was completed by English speaking patients in the United States only. LOCF was used for the Final visit analysis.
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 188 | 194 | 202
participants
  Baseline: Total | 182 | 188 | 196
  Baseline: Very Much Improved | 0 | 2 | 0
  Baseline: Much Improved | 6 | 6 | 3
  Baseline: Minimally Improved | 31 | 32 | 33
  Baseline: No Change | 126 | 134 | 148
  Baseline: Minimally Worse | 13 | 9 | 8
  Baseline: Much Worse | 3 | 5 | 4
  Baseline: Very Much Worse | 3 | 0 | 0
  Week 12: Total | 158 | 175 | 171
  Week 12: Very Much Improved | 13 | 22 | 28
  Week 12: Much Improved | 48 | 52 | 58
  Week 12: Minimally Improved | 53 | 59 | 42
  Week 12: No Change | 32 | 37 | 41
  Week 12: Minimally Worse | 6 | 4 | 2
  Week 12: Much Worse | 5 | 1 | 0
  Week 12: Very Much Worse | 1 | 0 | 0
  Final Visit: Total | 171 | 183 | 185
  Final Visit: Very Much Improved | 13 | 22 | 30
  Final Visit: Much Improved | 49 | 54 | 60
  Final Visit: Minimally Improved | 58 | 60 | 48
  Final Visit: No Change | 38 | 41 | 44
  Final Visit: Minimally Worse | 6 | 4 | 2
  Final Visit: Much Worse | 6 | 2 | 1
  Final Visit: Very Much Worse | 1 | 0 | 0

37. Secondary Outcome: Summary of Baseline, Week 12 and Final Visit Change in Bladder Symptoms on the Patient Global Impression Scale
Description: The patient global impression (PGI) scale assessed the change in bladder symptoms since the start of the study and was completed by the patient at Baseline and at Week 12/end of treatment. The degree of change was categorized as one of the following: 'Very much improved', 'Much improved', 'Minimally improved', 'No change', 'Minimally worse', 'Much worse', or 'Very much worse'.
Time Frame: Baseline and Week 12
Population: as for outcome 36
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 188 | 194 | 202
participants
  Baseline: Total | 188 | 194 | 202
  Baseline: Very Much Improved | 4 | 4 | 2
  Baseline: Much Improved | 14 | 15 | 12
  Baseline: Minimally Improved | 48 | 52 | 42
  Baseline: No Change | 105 | 105 | 124
  Baseline: Minimally Worse | 6 | 11 | 13
  Baseline: Much Worse | 5 | 5 | 9
  Baseline: Very Much Worse | 6 | 2 | 0
  Week 12: Total | 160 | 176 | 174
  Week 12: Very Much Improved | 18 | 23 | 37
  Week 12: Much Improved | 54 | 57 | 48
  Week 12: Minimally Improved | 49 | 57 | 45
  Week 12: No Change | 26 | 33 | 42
  Week 12: Minimally Worse | 5 | 5 | 1
  Week 12: Much Worse | 8 | 1 | 1
  Final Visit: Total | 173 | 185 | 188
  Final Visit: Very Much Improved | 18 | 23 | 39
  Final Visit: Much Improved | 54 | 60 | 51
  Final Visit: Minimally Improved | 52 | 57 | 49
  Final Visit: No Change | 35 | 36 | 45
  Final Visit: Minimally Worse | 6 | 7 | 1
  Final Visit: Much Worse | 8 | 2 | 3

38. Secondary Outcome: Summary of Baseline, Week 12 and Final Visit Change in Overall Condition on the Patient Global Impression Scale
Description: The patient global impression (PGI) scale assessed the change in the patient's overall condition since the start of the study and was completed by the patient at Baseline and at Week 12/end of treatment. The degree of change was categorized as one of the following: 'Very much improved', 'Much improved', 'Minimally improved', 'No change', 'Minimally worse', 'Much worse', or 'Very much worse'.
Time Frame: Baseline and Week 12
Population: as for outcome 36
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 188 | 194 | 202
participants
  Baseline: Total | 188 | 194 | 202
  Baseline: Very Much Improved | 3 | 5 | 2
  Baseline: Much Improved | 13 | 12 | 11
  Baseline: Minimally Improved | 46 | 47 | 41
  Baseline: No Change | 112 | 115 | 132
  Baseline: Minimally Worse | 6 | 12 | 11
  Baseline: Much Worse | 3 | 1 | 5
  Baseline: Very Much Worse | 5 | 2 | 0
  Week 12: Total | 160 | 176 | 174
  Week 12: Very Much Improved | 19 | 19 | 36
  Week 12: Much Improved | 47 | 60 | 51
  Week 12: Minimally Improved | 50 | 54 | 47
  Week 12: No Change | 33 | 39 | 38
  Week 12: Minimally Worse | 4 | 3 | 2
  Week 12: Much Worse | 7 | 1 | 0
  Final Visit: Total | 173 | 185 | 188
  Final Visit: Very Much Improved | 19 | 19 | 38
  Final Visit: Much Improved | 47 | 62 | 54
  Final Visit: Minimally Improved | 53 | 54 | 49
  Final Visit: No Change | 42 | 43 | 43
  Final Visit: Minimally Worse | 4 | 5 | 3
  Final Visit: Much Worse | 8 | 2 | 1

39. Secondary Outcome: Percentage of Participants With Improvement in Patient Perception of Bladder Condition (PPBC) at Week 12 and Final Visit
Description: The PPBC scale is a global assessment tool that asks patients to rate their impression of their current bladder condition on a 6-point scale from 1: 'Does not cause me any problems at all'; 2: 'Causes me some very minor problems'; 3: 'Causes me some minor problems'; 4: 'Causes me (some) moderate problems'; 5: 'Causes me severe problems' and 6: 'Causes me many severe problems'. Improvement was defined as at least a one point improvement from Baseline to post-baseline and a major improvement was defined as at least a two point improvement from Baseline to post-baseline in PPBC score.
Time Frame: Baseline and Week 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 postbaseline micturition measurement in the visit diary. The number of participants at each time point (N) only includes those with baseline and post-baseline values. LOCF was used for the Final Visit analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 415 | 410 | 426
percentage of participants
  Improvement: Week 12 [N=357; 381; 378] | 56.0 | 52.8 | 55.8
  Improvement: Final Visit [N=376; 391; 395] | 55.1 | 52.7 | 55.2
  Major Improvement: Week 12 [N=357; 381; 378] | 22.1 | 23.6 | 25.7
  Major Improvement: Final Visit [N=376; 391; 395] | 21.5 | 23.0 | 25.6

ADVERSE EVENTS:
Time Frame: Adverse events starting or worsening in the period from first double-blind study drug intake until 30 days after last double-blind study drug intake.
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg
Serious Adverse Events (participants affected / at risk) | 12/433 | 7/432 | 4/440
Other Adverse Events (participants affected / at risk) | 51/433 | 64/432 | 69/440
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=433) | Mirabegron 25 mg (N=432) | Mirabegron 50 mg (N=440)
Bronchitis acute (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Laparoscopy (Investigations) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Hemianopia homonymous (Nervous system disorders) | 1 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 1 | 0 | 0
Appendicectomy (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=433) | Mirabegron 25 mg (N=432) | Mirabegron 50 mg (N=440)
Hypertension (Vascular disorders) | 37 | 49 | 47
Nasopharyngitis (Infections and infestations) | 14 | 15 | 25

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.